CLINICAL TRIAL: NCT01882049
Title: Use of the REALIZE™ Adjustable Gastric Band (Model 2200-X) in Adolescents
Brief Title: Use of Adjustable Gastric Band in Adolescents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started due to funding issues
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE#G100290
Record Dates: First submitted 2012-11-20; First posted 2013-06-20 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: OBESITY
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Use of Realize gastric band (Ethicon) in adolescents for weight reduction
  Interventions: Device: REALIZE Gastric band (ETHICON)

INTERVENTIONS:
Device: REALIZE Gastric band (ETHICON) — Placement of gastric band around upper stomach

SUMMARY:
This study is to investigate the use the adjustable gastric band for the treatment of obesity in adolescents.

DETAILED DESCRIPTION:
Weight loss is related to the amount of energy or fuel obtained from the kinds and amounts of food eaten. When the amount of exercise and dieting uses less fuel than the amount taken in, the excess is stored as fat. The Adjustable Gastric Band used in this study is a tool to help the participant loose weight along with healthy eating, diet and exercise. This study involves minimally invasive laparoscopic surgery to place the adjustable band around the upper part of the stomach to make a smaller stomach or pouch about the size of a golf ball. One end of the band ends with a flat balloon that goes around the upper part of the stomach. The opening from this small stomach can be changed to allow more or less food into the intestine depending on the amount eaten and the amount of weight lost.

The other end of the of the band ends in a filling port through which saline solution is pumped with a needle through an attached tube to inflate or deflate the balloon. The filling port is attached to the wall of the abdomen under the skin. Because the flow of food is regulated by the band, most people feel full faster. This is how the appetite for food is controlled and the why the person is likely to eat less with the band in place.

Food is digested through the normal digestive process.

ELIGIBILITY:
Inclusion Criteria:

BMI: Female: ≥ 27 - ≥ 33 Male ≥ 26 - ≥ 30.5

Exclusion Criteria:

* •Hypertension: Systolic blood pressure (SBP) of 140 mm Hg

  * Hyperlipidemia: hyperlipidemia depends on
  * Obstructive Sleep Apnea:
  * Metabolic Syndrom: The presence of any three of the following: abdominal obesity - dimensons for children? triglycerides -cholesterol -
* fasting glucose
* blood pressure

  * overweight
  * Non-surgical means of weight reduction failure of
  * Significant psychopathology (absence of ) that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioral recommendations, as documented during screening assessment;
  * Agrees to refrain from any type of reconstructive surgery that would affect body weight such as abdominal lipoplasty or liposuction, mammoplasty, or removal of excess skin for three years following SAGB placement; and
  * Candidate for surgical weight loss intervention (i.e., meets accepted health criteria for major surgery.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | Monthly up to one year
  Reduction in percent of excess weight loss (%EWL).

CONTACTS AND LOCATIONS:
Overall Officials: Sayeed Ikrammudin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States